CLINICAL TRIAL: NCT05649488
Title: Evaluate the Safety and Efficacy of Intracoronary Lithotripsy Balloon Catheter and Intracoronary Lithotripsy Apparatus for Preconditioning of Coronary Calcified Lesions in a Prospective, Multi-center, Single-group Clinical Trial
Brief Title: Evaluate the Safety and Efficacy of Intracoronary Lithotripsy Balloon Catheter and Intracoronary Lithotripsy Apparatus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Bluesail Boyuan Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LFBY-202201
Record Dates: First submitted 2022-11-28; First posted 2022-12-14 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-12

CONDITIONS: Coronary Artery Disease; Intravascular Lithotripsy
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 184 patients were enrolled in the experimental group
  Interventions: Device: Intracoronary lithotripsy balloon catheter and Intracoronary lithotripsy apparatus
- Optical Coherence Tomography Subgroup (Other): 70 patients in the test group were enrolled in the OCT subgroup.
  Interventions: Device: Intracoronary lithotripsy balloon catheter and Intracoronary lithotripsy apparatus; Device: Dragonfly Opstar Imaging Catheter

INTERVENTIONS:
Device: Intracoronary lithotripsy balloon catheter and Intracoronary lithotripsy apparatus — Introduction: After the preparation, release the intracoronary lithotripsy balloon catheter to the area to be treated and release the shock wave pulse for treatment. After the balloon reaches the predetermined position, use angiography to lock the position and fill the balloon to 6 atm. After the shock wave pulse therapy, the balloon was expanded to 8 atm according to the balloon compliance table and lasted for 10s. After the treatment, unload the balloon pressure, wait for the blood flow to recover, and repeat the second treatment after an interval of one minute, two cycles, releasing a total of 20 shock wave pulses as a treatment cycle.
  Therapeutic apparatus specification: IVL-HVG-C01； Specifications of balloon catheter: C20012, C20015, C22512, C22515, C25012, C25015, C27512, C27515, C30012, C30015, C32512, C32515, C35012, C35015, C37512, C37515, C40012, C40015
Device: Dragonfly Opstar Imaging Catheter — OCT (optical coherence tomography) measurement using Dragonfly Opstar Imaging Catheter was performed in the OCT subgroup before or after the treatment of intracoronary lithotripsy balloon catheter and intracoronary lithotripsy therapeutic instrument, or after stent placement.
  Arms: Optical Coherence Tomography Subgroup

SUMMARY:
This is a prospective, multi-center, single-group target value clinical trial, which will be carried out in many clinical trial institutions in China. A total of 184 subjects (70 of them are OCT subgroups) are planned to be enrolled, all subjects were treated surgically with intracoronary lithotripsy using a balloon dilatation catheter and intracoronary lithotripsy apparatus after a single-group registration, clinical follow-up was carried out within 7 days after operation or before discharge, 1 month and 6 months after operation. The success rate of operation was taken as the main end point to verify the effectiveness of balloon dilatation catheter and intracoronary lithotripsy apparatus.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single-group target value clinical trial to recruit patients with coronary artery calcification, coronary artery calcification was pretreated with balloon dilatation catheter and intracoronary lithotripsy apparatus made by Shanghai Blusail Boyuan Medical Technology Co. , Ltd. , to verify the safety and efficacy of balloon dilatation catheter and intracoronary lithotripsy instrument for intravascular preconditioning of coronary artery calcification lesions. This trial will be carried out in many clinical trial institutions in China, and a total of 184 subjects (70 of them are OCT subgroups) are planned to be enrolled, all subjects were treated surgically with intracoronary lithotripsy using a balloon dilatation catheter and intracoronary lithotripsy apparatus after a single-group registration, clinical follow-up was carried out within 7 days after operation or before discharge, 1 month and 6 months after operation. In this study, the success rate of operation was taken as the main end point to verify the effectiveness of balloon dilatation catheter and intracoronary lithotripsy apparatus. A clinical summary report was issued for registration of the product 1 month after completion of postoperative follow-up, based on which a 6-month postoperative follow-up was performed to assess its safety. The secondary end points were angiographic success, device success, target lesion failure at 1 and 6 months, severe angiographic complications, MACE events at 1 and 6 months, serious adverse events and adverse events, and device defects. In the OCT Subgroup, the secondary end points were the minimum stent area (MSA), the minimum stent lumen diameter (MLD), the lumen acquired diameter, the lumen acquired area, and the lumen acquired rate of the immediate postoperative, the expansion rate of the stent, and the incomplete adherence rate of the stent beam.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, male or non-pregnant female.
2. Evidence of symptomatic ischemia, stable or unstable angina, or MI for more than 7 days.
3. Patients who can understand the purpose of the trial, voluntarily participate and sign the informed consent form, and are willing to undergo angiography, OCT and clinical follow-up.

Angiogram inclusion criteria

1. The target lesion was primary and in situ coronary artery disease.
2. Target lesion length ≤40 mm, target lesion reference vessel diameter 2.25-4.0 mm (visual inspection).
3. The target lesion diameter stenosis ≥70% or ≥50% (visual inspection) with evidence of ischemia.
4. Clear, high-density shadows can be seen both when the heart is beating and when it is not.
5. TIMI flow grade 3(allowing predilation) in the target vessel before use of the test equipment.
6. The target lesion was the only calcified lesion to be treated with the shock wave, and the non-target lesion needed to be treated successfully before the target lesion.
7. Suitable for patients undergoing metallic stent implantation

Exclusion Criteria:

1. Severe myocardial infarction occurred within 7 days before operation.
2. At the same time, the lesions were treated with rotational grinding or special balloon (chocolate balloon, nicked balloon, cutting balloon, double guide wire balloon, spinous process balloon, etc.).
3. NYHA Class III or IV.
4. Left ventricular ejection fraction <35% .
5. The target lesion was expected to be treated by fully biodegradable stent implantation, drug balloon dilatation and PTCA.
6. Uncontrollable severe hypertension (systolic blood pressure >180 mmHg or diastolic blood pressure > 110 mmHg).
7. Severe hepatic and renal impairment, transaminase more than 3 times the upper limit of normal, serum creatinine > 2.5 mg/dL (221 μmol/L), or chronic kidney failure requiring long-term dialysis.
8. Preoperative hemoglobin <100 g/l.
9. Platelet count <60×109/L.
10. Cerebral Stroke occurred within 6 months of enrollment, excluding transient ischemic attack (TIA) and lacunar infarction.
11. A history of active peptic ulcer or upper gastrointestinal bleeding within 6 months before enrollment.
12. Patients known to be allergic to heparin, contrast media, aspirin, clopidogrel and anesthetics.
13. Definite diagnosis of malignancy or life expectancy would be less than 12 months.
14. Participation in clinical trials of other drugs or medical devices that did not reach the primary end point.
15. The researchers judged that the patients had poor compliance and could not complete the study according to the protocol.

Angiographic exclusion criteria:

1. The target lesion was in the opening position (LAD, LCX or RCA, within 5 mm of the opening) or unprotected left main coronary artery.
2. Stents were implanted 10mm proximal or distal to the target lesion.
3. The target lesion had unprotected branch vessels more than 2.5mm in diameter.
4. The target lesion was distal to the saphenous vein or LIMA (Left internal mammary artery) /RIMA (Right internal mammary artery) bypass graft.
5. Existed an aneurysm within 10mm of the target lesion.
6. Angiography confirmed the presence of severe target lesion dissection (type D-F dissection (NHLBI classification) before the treatment of the Intracoronary lithotripsy balloon catheter and Intracoronary lithotripsy apparatus
7. The target lesion had definite thrombosis.
8. The researchers determined that the target lesion was unsuitable for vasodilation in patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
Operation success rate | During hospitalization (up to 7 days after operation)
  After successful stent placement, the residual stenosis in the stent is ≤ 30%, and there is no residual stenosis during hospitalization (up to 7 days after surgery at most) MACE event occurs

SECONDARY OUTCOMES:
Angiographic success rate (residual stenosis ≤ 30%) | Immediately after operation
  Efficacy endpoint
Incidence rate of MACE events 1 month and 6 months after operation | 6 months after operation
  Security endpoint
Target lesion failure (TLF) rate 1 month and 6 months after operation | 6 months after operation
  Security endpoint
Device success rate | 6 months after operation
  Security endpoint
Incidence of serious angiographic complications | 6 months after operation
  Security endpoint
Incidence rate of serious adverse events and adverse events | 6 months after operation
  Security endpoint
Incidence rate of device defects | 6 months after operation
  Security endpoint

OTHER OUTCOMES:
Minimum stent area (MSA) immediately after operation | Immediately after operation
  Secondary destination of OCT subgroup
Minimum stent lumen diameter (MLD) immediately after operation | Immediately after operation
  Secondary destination of OCT subgroup
Diameter of lumen obtained immediately after operation | Immediately after operation
  Secondary destination of OCT subgroup
Area of lumen obtained immediately after operation | Immediately after operation
  Secondary destination of OCT subgroup
Acquisition rate of lumen immediately after operation | Immediately after operation
  Secondary destination of OCT subgroup
Support expansion rate | Immediately after operation
  Secondary destination of OCT subgroup
Incomplete adherence rate of support beam | Immediately after operation
  Secondary destination of OCT subgroup

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, Ph.D, Principal Investigator — The General Hospital of Northern Theater Command
Locations (20):
- China (20):
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - the 980th Hospital of Chinese People's Liberation Army Joint Logistics Support Force, Shijiazhuang, Hebei
  - Fuwai Huazhong Cardiovascular Hospital, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - People's Hospital of Wuhan University, Wuhan, Hubei
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Second Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Cardiovascular Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Beijing Jishuitan Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Beijing Tsinghua Chang Gung Hospital, Beijing
  - Tianjin Chest Hospital, Tianjin
  - TEDA International Cardiovascular Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No